CLINICAL TRIAL: NCT07067866
Title: Weaning Approaches for Vasopressin in Sepsis - a Randomized Controlled Trial of Titrated Versus Abrupt Discontinuation During Stabilization of Septic Shock - WAVES Trial
Brief Title: Weaning Approaches for Vasopressin in Sepsis
Acronym: WAVES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Cássio Mallmann, Critical Care Physician, MS, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 83246724.1.0000.5530
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock
Keywords: vasopressin; septic shock; vasopressor weaning
MeSH Terms: conditions — Shock, Septic; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titrated group (Experimental): The titrated group will follow the vasopressin weaning protocol used in the DOVSS study (reduction of 0.01 U/min per hour).
  Interventions: Other: Titrated weaning of vasopressin.
- Abrupt group (Active Comparator): The abrupt group will discontinue the vasopressin infusion at the time of randomization, without dose titration.
  Interventions: Other: Abrupt weaning of vasopressin.

INTERVENTIONS:
Other: Titrated weaning of vasopressin. — The titrated group will follow the vasopressin weaning protocol used in the DOVSS study (reduction of 0.01 U/min per hour).
  Arms: Titrated group
Other: Abrupt weaning of vasopressin. — The abrupt group will discontinue the vasopressin infusion at the time of randomization, without dose titration.
  Arms: Abrupt group

SUMMARY:
In this study, we aim to evaluate the incidence of hypotension during vasopressin weaning by comparing two methods - titrated reduction versus abrupt withdrawal - through the conduct of a randomized clinical trial.

DETAILED DESCRIPTION:
Catecholamine infusions are usually tapered gradually in a titrated manner. However, little is known about how to manage adjunctive therapies such as vasopressin. While catecholamines have a short half-life (2-3 minutes), vasopressin's half-life ranges from 10 to 20 minutes. Although endogenous vasopressin levels are depleted in the early phase of shock, they are restored during recovery. Given its pharmacokinetic profile and the endogenous dynamics across different phases of shock, the optimal approach to vasopressin withdrawal - whether titrated or abrupt - remains unclear.

In 2021, a study was published comparing abrupt versus gradual vasopressin discontinuation. This was a retrospective observational study including 1,318 patients. Using ICU length of stay as the primary outcome, no significant difference was observed between groups (abrupt discontinuation: 7.9 days; gradual discontinuation: 7.3 days; p = 0.6). Similarly, there was no difference in the incidence of clinically significant hypotension (abrupt: 39.7%; gradual: 41.7%; p = 0.53). However, when stratifying patients based on whether catecholamine infusions were still ongoing at the time of vasopressin discontinuation, the results reversed in terms of ICU stay (abrupt: 9.2 days; gradual: 7.6 days), although this difference was not statistically significant (p = 0.24). In 2023, another retrospective observational study was published comparing abrupt versus gradual vasopressin withdrawal, including 74 patients. No difference was found in the incidence of clinically significant hypotension (abrupt: 57.1%; gradual: 52.3%; p = 0.68), nor in ICU length of stay. It is important to note, however, that in this cohort only patients who had already discontinued catecholamines prior to vasopressin withdrawal were included.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Admitted to the Intensive Care Unit
* Patients with vasopressor dependent sepsis
* Receiving combined norepinephrine and vasopressin therapy

Exclusion Criteria:

* Withdrawal/reduction of vasopressin related to a plan of treatment limitation or palliative care
* Withdrawal/reduction of vasopressin associated with the initiation of adrenaline or any other vasopressor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension within the first 24 hours | 24 hours
  Incidence of hypotension with clinical repercussions within the first 24 hours after titrated reduction or abrupt withdrawal of vasopressin.
  Definition of hypotension with clinical repercussions:
  mean arterial pressure < 60 mmHg, leading to:
  * administration of crystalloid/colloid bolus and/or
  * increase in norepinephrine dose and/or
  * reinitiation or increase in vasopressin dose.

SECONDARY OUTCOMES:
Hypotension stratified according to vasopressin duration | 24 hours
  Incidence of hypotension with clinical repercussions within the first 24 hours after titrated reduction or abrupt withdrawal of vasopressin, stratified according to vasopressin duration:
  < 48 hours
  ≥ 48 hours
  Definition of hypotension with clinical repercussions:
  mean arterial pressure < 60 mmHg, leading to:
  * administration of crystalloid/colloid bolus and/or
  * increase in norepinephrine dose and/or
  * reinitiation or increase in vasopressin dose.
Hypotension within the first hour | First hour
  Incidence of hypotension with clinical repercussions within the first hour after titrated reduction or abrupt withdrawal of vasopressin.
  Definition of hypotension with clinical repercussions:
  mean arterial pressure < 60 mmHg, leading to:
  * administration of crystalloid/colloid bolus and/or
  * increase in norepinephrine dose and/or
  * reinitiation or increase in vasopressin dose.
Vasopressor-free days | 7 days
  Number of days a patient is alive and free of vasopressor between randomization and day 7. Non-survivors will be considered to have zero vasopressor-free days.
Vasopressin-free days | 7 days
  Number of days a patient is alive and free of vasopressin between randomization and day 7. Non-survivors will be considered to have zero vasopressin-free days.
Renal replacement therapy | 7 days
  Initiation of hemodialysis between randomization and day 7, excluding chronic dialysis patients.
Cardiac arrhythmias | 7 days
  Incidence of arrhythmias with hemodynamic consequences between randomization and day 7, defined as hemodynamic deterioration requiring electrical or chemical cardioversion.
ICU-free days | 28 days
  Number of days a patient is alive and outside the ICU between randomization and day 28. Non-survivors will be considered to have zero ICU-free days.
Ischemic events | 28 days
  Occurrence of mesenteric ischemia, ischemic stroke, digital ischemia and acute coronary syndrome between randomization and day 28.
All-cause mortality | 28 days
  All-cause mortality within 28 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Cássio Mallmann, Critical Care Physician, MS, Principal Investigator — Hospital Nossa Senhora da Conceicao
Locations (1):
- Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Murata J, Buckley M, Lehn J, Agarwal SK, Stevenson B, Martinez B, MacLaren R. Incidence of Hypotension Associated With Two Different Vasopressin Discontinuation Strategies in the Recovery Phase of Septic Shock. J Pharm Pract. 2023 Aug;36(4):830-838. doi: 10.1177/08971900221078270. Epub 2022 Mar 25. PMID 35331049
- [Result] Lam SW, Sacha GL, Duggal A, Reddy AJ, Bauer SR. Abrupt Discontinuation Versus Down-Titration of Vasopressin in Patients Recovering from Septic Shock. Shock. 2021 Feb 1;55(2):210-214. doi: 10.1097/SHK.0000000000001609. PMID 32842024
- [Result] Der-Nigoghossian C, Hammond DA, Ammar MA. Narrative Review of Controversies Involving Vasopressin Use in Septic Shock and Practical Considerations. Ann Pharmacother. 2020 Jul;54(7):706-714. doi: 10.1177/1060028020901521. Epub 2020 Jan 20. PMID 31958982
- [Result] Jeon K, Song JU, Chung CR, Yang JH, Suh GY. Incidence of hypotension according to the discontinuation order of vasopressors in the management of septic shock: a prospective randomized trial (DOVSS). Crit Care. 2018 May 21;22(1):131. doi: 10.1186/s13054-018-2034-9. PMID 29784057
- [Result] Sacha GL, Lam SW, Duggal A, Torbic H, Reddy AJ, Bauer SR. Hypotension Risk Based on Vasoactive Agent Discontinuation Order in Patients in the Recovery Phase of Septic Shock. Pharmacotherapy. 2018 Mar;38(3):319-326. doi: 10.1002/phar.2082. Epub 2018 Feb 8. PMID 29328496
- [Result] Hammond DA, Painter JT, Meena N. Incidence of Clinically Significant Hypotension Stratified by Vasopressin Duration. J Intensive Care Med. 2019 Jan;34(1):77-78. doi: 10.1177/0885066617745809. No abstract available. PMID 30798676
- [Result] Landry DW, Levin HR, Gallant EM, Ashton RC Jr, Seo S, D'Alessandro D, Oz MC, Oliver JA. Vasopressin deficiency contributes to the vasodilation of septic shock. Circulation. 1997 Mar 4;95(5):1122-5. doi: 10.1161/01.cir.95.5.1122. PMID 9054839
- [Result] Bissell BD, Magee C, Moran P, Bastin MLT, Flannery AH. Hemodynamic Instability Secondary to Vasopressin Withdrawal in Septic Shock. J Intensive Care Med. 2019 Sep;34(9):761-765. doi: 10.1177/0885066617716396. Epub 2017 Jul 28. PMID 28750598
- [Result] Bauer SR, Aloi JJ, Ahrens CL, Yeh JY, Culver DA, Reddy AJ. Discontinuation of vasopressin before norepinephrine increases the incidence of hypotension in patients recovering from septic shock: a retrospective cohort study. J Crit Care. 2010 Jun;25(2):362.e7-362.e11. doi: 10.1016/j.jcrc.2009.10.005. PMID 19926252
- [Result] De Backer D, Deutschman CS, Hellman J, Myatra SN, Ostermann M, Prescott HC, Talmor D, Antonelli M, Pontes Azevedo LC, Bauer SR, Kissoon N, Loeches IM, Nunnally M, Tissieres P, Vieillard-Baron A, Coopersmith CM; Surviving Sepsis Campaign Research Committee. Surviving Sepsis Campaign Research Priorities 2023. Crit Care Med. 2024 Feb 1;52(2):268-296. doi: 10.1097/CCM.0000000000006135. Epub 2024 Jan 19. PMID 38240508
- [Result] Teboul JL, Duranteau J, Russell JA. Intensive care medicine in 2050: vasopressors in sepsis. Intensive Care Med. 2018 Jul;44(7):1130-1132. doi: 10.1007/s00134-017-4909-7. Epub 2017 Aug 31. No abstract available. PMID 28861671
- [Result] Leone M, Einav S, Antonucci E, Depret F, Lakbar I, Martin-Loeches I, Wieruszewski PM, Myatra SN, Khanna AK. Multimodal strategy to counteract vasodilation in septic shock. Anaesth Crit Care Pain Med. 2023 Jun;42(3):101193. doi: 10.1016/j.accpm.2023.101193. Epub 2023 Jan 5. PMID 36621622
- [Result] Hammond DA, Rech MA, Daley MJ, Devlin JW, Hodge EK, Kooda KJ, Lat I, Personett HA, Roberts R, Sacha G, Stollings JL, Swanson JM, Bauer SR. Perceptions regarding vasopressin use and practices in septic shock, and cost containment strategies. J Am Coll Clin Pharm. 2019 Jun;2(3):257-267. doi: 10.1002/jac5.1079. Epub 2019 Jan 24. PMID 38213315